CLINICAL TRIAL: NCT01036581
Title: Advanced Functional and Structural MRI Techniques for Neuropharmacological Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 999903380; 03-DA-N380
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-12-12

CONDITIONS: Drug Abuse; Nicotine Dependence
Keywords: Magnetic Resonance Imaging (MRI); Functional Brain Imaging; Magnetic Resonance Spectroscopy; Diffusion Tensor Imaging; Drug Abuse
MeSH Terms: conditions — Substance-Related Disorders; Tobacco Use Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MR Methodology Development and Evaluation (Experimental): Methodology development and evaluation consists of pulse sequence development, testing, and parameter optimization. For each method we develop or evaluate, we may recruit up to 40 participants to come in for up to 4 visits each. Each participant will be scanned for up to 2 sessions per visit, not to exceed 4 total scan hours per visit.
  Interventions: Device: Magnetom Prisma Fit 3T Scanner
- TMS-fMRI Experiment 1 (Experimental): To evaluate the relationship between BOLD activation and MEP and establish a BOLD activation marker of cortical excitability. Participants will start with a set of two short task-based EPI scans and anatomical scan. RMT will then be determined. Participants will undergo a single-pulse TMS-fMRI scan with stimulation intensities relative to the RMT over the motor cortex and/or the DLPFC. In total, six (6) intensities will be tested, 80% 100%, 105%, 110%, 115%, and 120% relative to the RMT. The fMRI design will be event-related. Each intensity (event type) will be presented 50 times. The order of the intensities will be randomized, and the inter-stimulus-interval (ISI) will range from 12s to 20s (centered at 16s plus random jittering in between, about 0.06Hz). The highest intensity of stimulation will be 120% RMT. EMG recordings in the corresponding hand muscle will be simultaneously acquired during the scan. Total approximate time required for this experiment is about 6-8 hours.
  Interventions: Device: MagPro X100 Magnetic Stimulator; Device: Transcranial Rotating Magnetic Stimulator
- TRPMS Experiment 1 (Experimental): To evaluate the prolonged effect of TPRMS on motor cortex excitability and help interpret and design subsequent experiments investigating the effect of TRPMS on BOLD signal. The experiment design consists of four groups, each group will include 10 participants (8 completers/group). For TRPMS stimulation sessions, our test conditions will be a 10 stimuli-session (approximately 2min), 50 stimuli-session (approximately 7min), 100 stimuli-session (approximately 14min), and 150 stimuli-session (20min) for each of the four groups, respectively. Therefore, the outcome will be measured with the spontaneous motor unit potentials (sMUPs) in the contralateral abductor pollicis brevis muscle (APB). After the stimulation session, we will measure sMUPs continuously for another 20min to observe the prolonged effect of the TRPMS stimulation and to compare these four conditions. The total approximate time required for this experiment is about 2-2.5 hours.
  Interventions: Device: Transcranial Rotating Magnetic Stimulator
- TRPMS Experiment 2 (Experimental): To evaluate cortical excitability changes caused by TRPMS measured with simultaneous TMS-fMRI. Participants will undergo a baseline TMS/fMRI session to get a measurement of baseline cortical excitability in the form of single-pulse TMS induced BOLD activation and determine motor hot-spot and RMT. We will then conduct an event-related single-pulse TMS/fMRI session with TMS stimulus at 120% RMT, 50 events with jittered inter-stimulus-interval (ISI) averaging 16s. Simultaneous EMG recording will be gathered from the corresponding hand muscle. Next we will use TRPMS to stimulate the left motor cortex over the hot-spot : 20-min application of TRPMS, 100ms duration, 0.2Hz (one stimulus every 5s), total 240 stimuli. Then we will evaluate the modulatory effect of the TRPMS stimulation via a second TMS/fMRI session with a similar procedure as the baseline session using the RMT determined at baseline. Total time for this experiment is about 5-6 hours.
  Interventions: Device: MagPro X100 Magnetic Stimulator; Device: Transcranial Rotating Magnetic Stimulator

INTERVENTIONS:
Device: MagPro X100 Magnetic Stimulator — Concurrent TMS-MRI acquisition allows us to investigate the acute effects of induced brain activity on BOLD signal and evaluate interference of the TMS pulse with the BOLD signal measurement.
  Arms: TMS-fMRI Experiment 1; TRPMS Experiment 2
Device: Transcranial Rotating Magnetic Stimulator — Participants will undergo transcranial rapid rotating permanent magnetic stimulation (TRPMS), with the aim of evaluating the prolonged effect of TRPMS on motor cortex excitability. In another experiment, participants will undergo TRPMS with the aim of evaluating cortical excitability changes with TRPMS. These experiments will help interpret subsequent experiments investigating the effect of TRPMS on BOLD signal.
  Arms: TMS-fMRI Experiment 1; TRPMS Experiment 1; TRPMS Experiment 2
Device: Magnetom Prisma Fit 3T Scanner — Type: MRI Name: Magnetom Prisma Fit 3T Scanner (Siemens) Description: Functional and structural magnetic resonance imaging techniques are used for noninvasive mapping of brain physiology and pathology and to develop advanced magnetic resonance imaging and spectroscopy (MRI and MRS) techniques for neuroimaging studies related to addiction.
  Arms: MR Methodology Development and Evaluation

SUMMARY:
Background:

- Functional and structural magnetic resonance imaging (MRI) techniques have allowed researchers to map and study how the brain works when at rest and when engaged in specific tasks. MRI scans have provided more information about how drugs affect the brain, and about how drug addiction changes the brain and influences behavior, mood, and thinking processes. To better understand the underlying mechanism of drug addiction and to develop strategies for more effective treatment, researchers are interested in developing new MRI techniques to study the effects of addiction on the brain.

Objectives:

- To develop new functional and structural MRI techniques, and to evaluate their potential use in brain imaging studies related to addiction.

Eligibility:

* Individuals between 18 and 80 years of age.
* Participants may be smokers or nonsmokers, and may use drugs or not use drugs.

Design:

* During the initial screening, participants will complete questionnaires about family and personal history, drug use, and other information as required by the researchers. Participants who will be asked to complete tasks during the MRI scan will be shown how to perform these tasks before the scanning session.
* Before each study session, participants may be asked to complete some or all of the following: questions about their drug use during the last week, a breathalyzer test, a urine drug-use assessment, a urine pregnancy test, or a measure of carbon monoxide. Participants will also provide blood samples before the start of the scan.
* For each scanning session, participants will have an MRI scan that will last approximately 2 hours.
* MRI scans may include specific tasks to be performed during the scan, or an experiment that studies the brain's response to carbon dioxide....

DETAILED DESCRIPTION:
Objective:

Functional and structural magnetic resonance imaging techniques have proven essential for noninvasive mapping of brain physiology and pathology. The primary objective of this protocol is to develop advanced magnetic resonance imaging and spectroscopy (MRI and MRS) techniques for neuroimaging studies related to addiction. These neuroimaging techniques will be used in other studies to better understand the underlying mechanism of drug addiction and to potentially develop strategies for more effective treatment.

Study population:

Healthy controls and drug users will participate in the study. Technical developments of MRI/MRS will be performed on healthy controls, while the evaluation of the applicability of these techniques to addiction related neuroimaging studies will be performed using drug users and healthy controls.

Design:

Based on the fundamental principle of the biophysical transduction of physiological signals to magnetic resonance (MR) imaging and spectroscopic signals, advanced techniques will be developed to measure the activity, metabolism, structure, and biochemistry of the brain. The development of these techniques typically includes the following steps: 1) proof-of-concept computer simulations, 2) implementation of the imaging concept with an MRI scanner and phantoms, 3) feasibility testing on control subjects, and 4) evaluation of the sensitivity and specificity of these techniques in detecting functional changes modulated by task performance, CO2 (5%)administration, or non-invasive neuromodulation techniques (e.g.: transcranial magnetic stimulation (TMS), and transcranial rotating permanent magnet stimulation (TRPMS), 5) evaluation of these techniques in detecting functional and/or structural alterations of the brain related to a specific disease.

Outcome measures:

Advanced neuroimaging techniques developed from this protocol will demonstrate the ability to distinguish between drug using and control populations. Successful techniques will then be incorporated into hypothesis driven studies in the Neuroimaging Research Branch at NIDA-IRP. These techniques will also be useful, through publications and technology transfer, to the entire neuroimaging society.

ELIGIBILITY:
* Subjects must be between the ages of 18-80, be generally healthy and male or non-pregnant female. Smokers, non-smokers, drug using and non-drug using populations will participate in this study.

INCLUSION CRITERIA:

General:

* Male and non-pregnant female adults between the ages of 18-80.
* All subjects must be able to provide informed consent.

EXCLUSION CRITERIA:

Subjects will be excluded if they:

* Are pregnant. Urine pregnancy tests will be performed on all female volunteers of child-bearing potential before each experimental session.
* Are unable to undergo MRI scanning due to implanted metallic devices (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips or other implanted metal parts including Copper 7 IUD) or claustrophobia.
* Have major medical illnesses severe enough to impact data being gathered. Potential exclusions may include a history of chronic uncontrolled hypertension, diabetes, HIV, or other clinically significant medical conditions that may alter the signal being measured.
* Have current major psychiatric disorders to include, but not limited to, mood, anxiety, psychotic disorders.
* Have neurological illnesses severe enough to impact data being gathered. Potential exclusions may include seizure disorders, migraine, multiple sclerosis, movement disorders, or history of significant head trauma, CVA, or CNS tumor. The MAI will assess the severity in relation to the potential impact on data.
* Are non-English speaking. Justification: There is no direct benefit to participants in this study, and some of the study procedures involve more than minimal risk. To include non-English speakers, we would have to translate the consent and other study documents and hire and train bilingual staff, which would require resources that we do not have and could not justify given the small sample size for each experiment. Additionally, the data integrity of some of the cognitive tasks and standardized questionnaires used in this study would be compromised as they have only been validated in English. Most importantly, ongoing communication regarding safety procedures is necessary when participants are undergoing MRI and TMS/TRPMS procedures. The inability to effectively communicate MRI and TMS/TRPMS safety procedures could compromise the safety of non-English speaking participants.
* Are cognitively impaired, as assessed by the consent quiz and medical history. A validated IQ test such as the WASI or Shipley-2 may also be considered. Justification: Cognitive impairment and learning disabilities are associated with alterations in brain regions used to accomplish tasks, and, therefore, may introduce significant variably into the data. Cognitive impairment may affect one s ability to give informed consent.

Subjects to be considered for Non-Invasive Brain Stimulation (NIBS) will also be excluded if they:

-Are unable to safely undergo a NIBS procedure as assessed by a TMS safety screening form.

Additional information will be gathered during screening for some experiments. As the purpose of this protocol is to develop imaging techniques, this information will be gathered as needed, depending on the phase of development and specific technique requirements. Based on the scientific and medical requirements of the particular experiment, participants may also be assessed for:

* age (some experiments may want to target a particular age range. For example, cognitive tasks generally exclude participants over 60, an age when cognitive issues tend to become more commonplace)
* left-handedness (if desired for a particular task)
* color-blindness (if using a task requiring color discrimination)
* drug use diagnosis
* use of psychoactive or vascularly active medications (if a functional fMRI technique that is sensitive to hemodynamic changes is being used)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2003-10-24 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
To develop a simultaneous perfusion and BOLD imaging technique with improved functional contrasts and reduced susceptibility artifacts for determination of CMRO2 during brain activation | at each visit
  perfusion/BOLD imaging data
To develop efficient methods to reduce image artifacts caused by susceptibility-induced field inhomogeneity and head motion, and therefore to improve reliability and sensitivity of functional imaging | at each visit
  MRI scan data
To develop an imaging technique to identify fiber crossing in the brain based on high-angular resolution measurements of apparent diffusion coefficient (ADC), and subsequently to develop improved fiber tracking techniques to delineate neuronal p... | at each visit
  MRI scan data
To develop MRS techniques that are able to reliably measure metabolite and neurotransmitter concentrations in the brain at 3 Tesla, and to evaluate their feasibility and efficacy in drug addiction studies | at each visit
  MRS data from MRI scans
To integrate genetic analysis with morphological and functional measurement of the amygdala, hippocampus, and other regions, which may help to account for some of the noise in these measurements | at each visit
  MRI scan data and blood samples collected in 380 or 457 (NRB genetics protocol).
To assess effects of neuromodulation techniques, such as TMS and TRPMS, on brain activity and relevant MRI signals | at each visit
  MRI scan data; spontaneous motor unit potentials (sMUPs) in the contralateral abductor pollicis brevis muscle (APB)

CONTACTS AND LOCATIONS:
Overall Officials: Yihong Yang, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share IPD for this protocol with properly administered databases and/or with collaborators with whom proper data sharing agreements are in place (please see summary of data sharing agreements in the protocol); Not all plan details have been finalized. We have not yet finalized decisions on types of supporting information that will be shared, IPD Sharing Time Frame, or IPD Sharing Access Criteria for all agreements or databases.